CLINICAL TRIAL: NCT05059821
Title: Phase I Clinical Trial of Alfa-Fetoprotein,Glypican-3 Based Personalized Cancer Vaccine in Egyptian Patients With Hepatocellular Carcinoma: Pilot Study
Brief Title: Personalized Cancer Vaccine in Egyptian Cancer Patients
Acronym: PROVE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: zeinab ahmed yousif hasan ashour (Other)
Responsible Party: Sponsor-Investigator, zeinab ahmed yousif hasan ashour, Professor of Internal Medicine, Allergy and clinical immunology unit, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P109g/2019-2021
Record Dates: First submitted 2021-05-11; First posted 2021-09-28 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Peptide vaccine, Heat shock protein 70, Monocytes
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Personalized peptide based vaccine with autologous heat shock protein 70 and autologous activated monocytes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Personalized Cancer Vaccine (Experimental): Patients with recurrent HCC after surgical resection and refractory to available line of treatment will receive Personalized peptide based vaccine with autologous heat shock protein 70 and autologous activated monocytes
  Interventions: Biological: Peptide cancer vaccine

INTERVENTIONS:
Biological: Peptide cancer vaccine — Vaccine content are personalized peptides vaccine separated from each patients own tumor cells, autologous heat shock protein 70 separated from tumor cells and autologous activated monocytes that administered subcutaneously monthly for six months

SUMMARY:
Evaluate safety and immunogenicity of peptide cancer vaccine in patients with hepatocellular carcinoma (HCC) who developed recurrence after surgical resection and refractory to the available institutional standard of care lines of treatment .

DETAILED DESCRIPTION:
Ten patients with hepatocellular carcinoma (HCC) who developed recurrence after surgical resection are refractory to the available institutional standard of care lines of treatment will be recruited to received the peptide cancer vaccine.

Tumour antigen peptides will be identified and separated from each patient and then reinjected with an adjuvant (autologous activated monocytes with autologous tumour derived heat shock protein 70) by subcutaneous route monthly for 6 months preceded by 300 mg cyclophosphamide one week before start of the vaccine.

A follow up for all cases will be performed clinically, laboratorial, and immunologically for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who developed recurrence of HCC after surgical resection .
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group performance status (ECOG) of 0-2 .
4. Patient with radiologically or pathologically confirmed hepatocellular carcinoma.
5. Patients who had been treated with surgical approach as per our (Ain Shams University) institute protocols and developed recurrence after surgery. They were either intolerant to the institute protocol of treatment or showed unresponsiveness of their disease after treatment.
6. Child-Pugh class A or B .
7. LAB values:

   Hemoglobin (≥ 8 g/dl), platelets (≥ 50,000/µl), leukocytes (≥ 2,500/µl), neutrophils (≥ 1,000/µl), lymphocytes (≥ 500/µl) Liver function: serum bilirubin (< 3 x ULN), Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) (< 5 x ULN) Renal function: serum creatinine (< 1.5 x ULN)
8. Patient has not received any antineoplastic chemotherapy, immunotherapy, or radiotherapy for the four weeks prior to the start of study treatment.
9. Pregnancy test should be negative at the first dose of study treatment in fertile females. (Female patients who are not post-menopausal or surgically sterile should use a highly effective method of birth control from the date of signing the consent to the last follow up visit. Pregnancy test should be negative at the first dose of study treatment.)
10. Written informed consent .

Exclusion Criteria:

1. Patients receiving continuous systemic steroid treatment within the last 4 weeks prior to start of study treatment (The use of inhaled and nasally applied steroids, as well as topical steroids outside the vaccination area are permitted)
2. Patients receiving systemic immunotherapy or immunosuppressant medication other than steroids within the last 4 weeks prior to start of study treatment.
3. Patients with a history or evidence of systemic autoimmune disease.
4. Active second malignancy or a prior malignancy within the past 12 months.
5. Acute active infections requiring oral or intravenous antibiotics, antiviral or antifungal therapy within 1 week before the start of study treatment [Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infections are permitted; direct-acting antivirals may be administered when medically indicated].
6. Any other acute medical condition that may compromise patient's safety or the activity of the studied vaccine treatment.
7. Any other concurrent severe or uncontrolled chronic disease such as uncontrolled non-malignant liver, renal or lung disease, or decompensated cardiac failure or coronary insufficiency.
8. Administration of a live, attenuated vaccine within 4 weeks before randomization
9. Known previous major hypersensitivity reactions.
10. History of human immunodeficiency virus (HIV)
11. Evidence of current alcohol or drug abuse
12. Women who are pregnant or who are breast feeding
13. Medical or mental impairments that may limit participation in the study as judged by the investigators disease specialist.
14. History of organ allograft.
15. History of splenectomy.
16. Psychiatric illness or known social situation that would preclude study compliance.
17. Encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety of the personalized cancer vaccine | 4 weeks
  Percentage of patients who developed adverse events (AEs)
Assessment of immunological response | 12 weeks
  Percentage of change in CD20 +B-cells, CD16+CD56+NK cells,CD4 + cells,CD8+ cells,CD25+regulatory cells

SECONDARY OUTCOMES:
Progression free survival and overall survival time | 144 week
  Progression free survival (PFS) time and overall survival (OS)time will be analysed using the Kaplan-Meier estimation method and log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab A Ashour, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams Research Institute- Clinical Research Center (MASRI-CRC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No